CLINICAL TRIAL: NCT05705128
Title: Comparison Between Effect of Addition of Dexamethasone and Dexmedetomidine in Combination With Bupivacaine for Pain Relief After Shoulder Arthroscopic Surgeries
Brief Title: Dexmedetomidine in Postoperative Analgesia
Acronym: Any
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Abdelsabour, lecturer, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Assiut anesthesia g35
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-11

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone group (Active Comparator): patients will receive dexamethasone with bupivacaine before general anaesthesia
  Interventions: Drug: Dexmedetomidine
- dexmedetomidine group (Active Comparator): patients will receive dexemedetomidine with bupivacaine before general anaesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be given with bupivaciane for postoperative pain control

SUMMARY:
There is a high incidence reaching up to 45%; of severe intraoperative and postoperative pain associated with arthroscopic shoulder surgery, which is often significant enough to interfere with initial recovery and rehabilitation.Various peripheral nerve blocks have been used to reduce intraoperative anesthetic requirements to improve rapid recovery and reduce postoperative pain.

DETAILED DESCRIPTION:
Recently, the Combined suprascapular nerve block and axillary nerve block (SSNB+ANB) was proposed to provide anesthesia and postoperative analgesia for shoulder surgery as a safe alternative to ISB.most of the nerve supply from C5 and C6 nerve roots are carried by suprascapular and the axillary nerves. These two peripheral nerves are responsible for the majority of the sensory innervation of the shoulder.

Dexamethasone is a glucocorticoid that is commonly used to decrease the body's inflammatory response. Doses of 1, 2, 4, and 8 mg have been used as an adjuvant in interscalene, supraclavicular, ankle, and brachial plexus blocks . However, when dexamethasone is used as an adjuvant in a PNB, the specific mechanism of action is unknown . Dexamethasone may produce extended analgesia through vasoconstriction and reduced absorption of local anesthetic or through "direct action on the nerve cell to reduce neural discharge" .

Despite having an unknown mechanism, a Cochrane review of 35 trials of 2702 participants determined that perineural dexamethasone adjuvant increased sensory block 6.7 hours (95% confidence interval) in comparison to a placebo . Similarly, intravenous dexamethasone increased sensory block 6.2 hours in comparison Dexmedetomidine is a highly selective and potent central alpha-2 adrenergic receptor agonist. Administration of this adjuvant in miscellaneous methods has received considerable attention in recent years. Due to its analgesic and sedative effects, besides the lack of any respiratory-sparing effects, administration of this adjuvant has been effective in reducing the need for opioids in the perioperative period and may even result in cooperative sedation . Given the sympatholytic effects of dexmedetomidine (hypotension and bradycardia), in addition to oversedation, especially when administered intravenously or at high doses, caution must be taken in administering this drug, especially in elderly patients.

The neuraxial administration of dexmedetomidine has nociceptive effects on somatic and visceral pains . It also reduces postoperative pain and prolongs analgesia, although there is a risk of bradycardia. Various doses of dexmedetomidine, along with a number of analgesic drugs, have been used in many studies. However, the exact dose of dexmedetomidine, as an adjuvant drug administered along with other intravenous drugs in the perioperative period, has been controversial.

The proposed mechanism for perineural dexmedetomidine in PNBs as first studied in rat models is similar to that of clonidine, which relies not on alpha-2 agonism mechanism, but instead blocks hyperpolarization-activated Ih cation currents and causes vasoconstriction for prolonged analgesia . Perineural dexmedetomidine adjunct use is off-label, and proper risk-benefit analysis, especially in patients where bradycardia and hypotension would be concerning, would be necessary before even more widespread use of dexmedetomidine in PNBs can be expected .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective shoulder arthroscopy under general anesthesia

Exclusion Criteria:

* Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis).
* Altered conscious level.
* Pregnancy. .Body mass index (BMI > 35).
* Patients who have difficulty understanding the study protocol
* Patients who have any known contraindication to study medications
* Patient refusal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
numerical rating pain scale | 24 hours
  graded from 0 to 10 (0 = no pain, 10 = the worst possible pain)

SECONDARY OUTCOMES:
complications | 24 hours
  postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abdelsabour, lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No